CLINICAL TRIAL: NCT01425684
Title: Brain Circuits in Schizophrenia and Smoking
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, MPRC, Associate Professor, University of Maryland, Baltimore
Other Study IDs: HP-00045716; R01DA027680 (NIH)
Record Dates: First submitted 2011-08-28; First posted 2011-08-30 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: MRI; Smoking; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Whole Blood
  * Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- schizophrenia: smokers and nonsmokers
- control: smokers and nonsmokers

SUMMARY:
The principle aim of the project is to identify the key brain circuits associated with smoking and especially smoking in high risk population. The investigators hope that the study will provide concrete biomarkers for new therapeutic development and ultimately reducing the smoking related health burden.

DETAILED DESCRIPTION:
There are several studies and hypotheses to be tested. This project includes (1) a cross-sectional study design that measures brain imaging, smoking, clinical diagnosis and symptoms, cognitive functional assessments, distress tolerance, and genetic information, which is also the baseline for the longitudinal study; and (2) a longitudinal study design for smoking cessation option for 1 year in some smokers and a longitudinal follow-up for all available subjects.

During the baseline portion of the study, subjects are expected to complete clinical symptom assessments, a computer challenge task to measure distress tolerance, MRI scan, role-play test to measure cognitive and functional abilities, and blood draw. Subjects who are eligible will participate in the longitudinal follow-up study where the research team will call subjects regularly regarding smoking related information (smoking risk and treatment options).

ELIGIBILITY:
Inclusion Criteria:

* Male and Female between ages 12-above (clinical assessments and blood draw only above 62)
* Ability to give written assent (age below 18)
* Ability to give written informed consent (age 18 or above)
* Individuals fulfilled other criteria but over age 62, with major medical illnesses, significant alcohol or other drug use, or unable to undergo MRI may participate in clinical assessments and blood draw if his/her participation forms a family unit (i.e., if at least one of the family member has participated).
* Subjects above age 62 will not participate in MRI measurements although they may still participate in clinical assessments and blood draw.

Exclusion Criteria:

* Inability to sign informed consent/assent
* For patient participants, Evaluation to Sign Consent (ESC) below 10.
* Any major medical illnesses that may affect normal brain functioning. Examples of these conditions include, but not limited to, stroke, repeated seizure, history of significant head trauma, CNS infection or tumor, other significant brain neurological conditions.
* Significant alcohol or other drug use (substance dependence within 6 months or substance abuse within 1 month) other than nicotine or marijuana dependence.
* Woman who are pregnant (child-bearing potential but not on contraceptive and missing menstrual period; or by self-report; or by positive urine pregnancy test before MRI)
* Can not refrain from using alcohol and/or marijuana 24 hours or more prior to experiments.
* For MRI, unable to undergo MRI scanning due to metallic devices or objects (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts) or claustrophobic to the scanner

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Smokers, nonsmokers, schizophrenia patients, family members
Sampling Method: Non-Probability Sample
Enrollment: 837 (Actual)
Dates: Start 2010-12-20 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Nicotine addiction severity is associated with abnormal functional connectivity as measured by fMRI,compared with nonsmokers.Schizophrenia pts are assoc with add'l functional connectivity impairment compared with controls | 12-15 hours

SECONDARY OUTCOMES:
Symptom and Cognition rating | 1-2 hours

CONTACTS AND LOCATIONS:
Overall Officials: L.Elliot Hong, M.D., Principal Investigator — Maryland Psychiatric Research Center, Department of Psychiatry, University of Maryland School of Medicine
Locations (1):
- Maryland Psychiatric Research Center, Department of Psychiatry, University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No